CLINICAL TRIAL: NCT07395765
Title: Acute Serum Brain-Derived Neurotrophic Factor (BDNF) and Executive Function Responses to Touch-Limited vs Free-Play 4v4 Small-Sided Games in Male Soccer Players
Brief Title: Comparing Touch-Limited and Free-Play 4v4 Small-Sided Games (SSGs)
Acronym: TOUCH-BDNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, serkan pancar, Assoc. Prof., Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21.13
Record Dates: First submitted 2026-02-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: BDNF; Small Side Game; Football Players
Keywords: BDNF; Lactate; Cognitive Performance; SSG

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSGf (Experimental)
  Interventions: Behavioral: SSGf
- SSGr (Experimental)
  Interventions: Behavioral: SSGr

INTERVENTIONS:
Behavioral: SSGf — The SSGf was free-flowing without imposed constraints, such as touch limitations, mandatory passing, or predefined scoring conditions.
  Other Names: Small Sided Games Free
  Arms: SSGf
Behavioral: SSGr — The only difference from the free-play condition was limiting the number of ball touches. Accordingly, each time players received the ball, they were required to release it by the second touch at the latest (e.g., via a pass or shot). In the event of a violation of this two-touch rule (i.e., >2 touches), possession was immediately awarded to the opposing team to preserve the continuity of play.
  Other Names: Small Sided Games Rules
  Arms: SSGr

SUMMARY:
This study aimed to compare acute serum BDNF and cognitive performance following touch-limited versus free-play 4v4 small-sided games (SSGs) in male soccer players.

This randomized crossover controlled trial aimed to examine the acute effects of touch-limited (SSGr) vs free-play (SSGf) 4v4 SSGs on serum brain-derived neurotrophic factor (BDNF), blood lactate levels and executive function performance in male soccer players. All participants completed the two conditions in a randomized and counterbalanced manner. To ensure balanced exposure, they were assigned to one of two groups (n=16), each following a distinct condition. A seven-day interval separated each session to reduce residual physiological or cognitive effects. The trial protocol was developed in line with Consolidated Standards of Reporting Trials guidelines, including for within-subject designs and non-pharmacological interventions. Participants were blinded to the study hypothesis.

Teams were formed based on the coach's assessment of the players' technical, tactical, and physical abilities. To minimize differences in player's maximum oxygen consumption (VO2 max) level estimated from the 30-15 Intermittent Fitness Test (30-15 IFT) were also taken into account.

The SSG sessions were conducted at 10.00-12.00 to have similar chronobiological characteristics on a natural grass pitch during the off-season period under the supervision of A-licenced coaches to ensure consistency and adherence to protocol. All players continued their routine off-season training program, which involved three training sessions (strength, aerobic activity, aerobic running) per week. Players were advised to avoid strenuous exercise within 48 h, be prohibited from drinking alcohol or coffee within 24 h, and have at least 7-8 h of sleep before the intervention. During this study, the players were instructed to maintain their dietary habits and general lifestyle.

During the first visit, participants' resting heart rate was recorded. Then body weight and body fat percentage were assessed using bioelectrical impedance analysis. To mitigate potential learning effects, all participants underwent a familiarization session with Stroop Test. Finally, participants performed 30-15 IFT to determine aerobic capacity, and peak heart rate.

During the two subsequent visits, each participant completed both SSGr and SSGf sessions, with one session (SSGr or SSGf) completed during visit 2 and the other during visit 3. The half of the participants completed SSGr first and the other half completed the SSGf first.

Blood samples were collected and cognitive performance tests were conducted before and after each training session. The heart rate was monitored throughout each session. Additionally, following each exercise session, rating scale mental effort scores were used to assess the players' psychophysiological responses. Water intake was permitted during all the recovery periods throughout the training sessions.

Each exercise session began with a standardized 10-minute warm-up, including light jogging, dynamic stretching, and soccer-specific movement preparation drills with and without the ball. All exercise sessions lasted 40 minutes in total, consisting of a 10-minute standardized warm-up, 24 minutes of exercise, and a 5-minute recovery period.

In this study, we conducted 4v4 SSG to foster environments recommended by studies suggesting that game formats with fewer players may offer a more cognitively demanding structure, including creativity, exploratory behaviors, and decision-making challenges for players. The SSGs with mini-goals were played on a 30 × 24 m pitch (720 m²), with dimensions set to provide a comparable relative area per player (90 m²). The duration of the SSG was carefully standardized, consisting of four 4 min bouts with 3 min passive recovery intervals between bouts. During recovery, players went to the sideline for ad libitum rehydration and returned to their positions in walking speed. These movements were excluded from analysis as they are not representative of match play. Across all experimental conditions, participants were encouraged to maximize the number of goals scored to foster a competitive environment and sustain a high level of effort. Players were instructed to exert maximal effort during gameplay and received verbal encouragement, which excluded feedback on their technical and tactical performance. To ensure uninterrupted play and maximize effective playing time, multiple balls were placed along the sidelines, and two coaches stationed around the field promptly provided replacement balls when required. The SSGf was free-flowing without imposed constraints, such as touch limitations, mandatory passing, or predefined scoring conditions. In the SSGr, the only difference from the free-play condition was limiting the number of ball touches. Accordingly, each time players received the ball, they were required to release it by the second touch at the latest.

ELIGIBILITY:
Inclusion Criteria:

* Semi-professional male soccer players with ≥10 years of soccer experience
* Aged between 18 and 25 years
* No known medical condition that prevents participation in exercise
* No recent use of medications or supplements that could enhance anaerobic or aerobic performance
* No recent severe lower-extremity injury (>12 months)

Exclusion Criteria:

* Experiencing any discomfort before, during, or after exercise
* History of alcohol or substance addiction
* Any other condition or factor that may prevent full participation in the study protocol
* Being a goalkeeper

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants are eligible to participate in this study based on biological sex.
Enrollment: 32 (Actual)
Dates: Start 2025-07-23 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
BDNF | • Baseline, Immediately After Exercise (Day 1)
  BDNF levels were measured using a Sunred Brand Enzyme-Linked İmmunosorbent Assay (ELISA) kit from blood samples taken baseline and after exercise, and the results were reported in ng/mL units.
Lactate | • Baseline, Immediately After Exercise (Day 1)
  Lactate levels were measured in millimoles per liter (mmol/L) from capillary/venous blood samples taken before and after exercise using a lactate analyzer.
Stroop Test | • Baseline, immediately after exercise (Day 1)
  The Stroop Test is a widely used neuropsychological assessment tool to evaluate selective attention, inhibitory control, processing speed, and executive function under cognitive interference.
  The Congruent condition measures baseline color-naming speed by requiring participants to respond to stimuli in which the color word matches the ink color. Completion time (or reaction time) and errors were recorded.
  The Incongruent condition measures inhibitory control and interference resolution by requiring participants to name the ink color while ignoring a conflicting color word. Completion time (or reaction time) and errors were recorded.
  Performance was evaluated using (i) condition-specific completion/reaction times and error counts and (ii) the Stroop interference score, calculated as the difference between conditions (Incongruent - Congruent) for time (and/or errors). Lower interference values reflect better inhibitory control and interference resolution, whereas higher va
Rating Scale Mental Effort | • Immediately After Exercise (Day 1)
  RSME (Rating Scale Mental Effort) is a single-item measure scored on a 0-150 continuum. Immediately after each session, participants indicate their perceived mental effort by marking a 150-mm visual analogue line anchored with verbal descriptors; the distance from the origin is measured in millimeters and recorded as the RSME score (0-150). Higher scores reflect greater perceived mental effort (i.e., a higher cognitive/mental demand imposed by the session).
Feeling Scale | • Baseline, Immediately After Exercise (Day 1),
  The Feeling Scale (FS) is a single-item measure used to assess affective valence during exercise and is scored on an 11-point scale ranging from -5 to +5. Participants select the value that best reflects how they feel at a given time point (e.g., during or immediately after exercise), where -5 indicates "very bad," 0 represents a neutral feeling, and +5 indicates "very good." Higher scores denote more positive affective responses, whereas lower scores reflect more negative affective states.

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality concerns arising from the small sample size and the collection of sensitive biomarker and performance-related measures. The combination of these variables increases the risk of participant re-identification through data triangulation, even after anonymization. To protect participant privacy and ensure compliance with ethical approval and data protection regulations, individual-level data will therefore not be made publicly available. Only aggregated results are reported.